CLINICAL TRIAL: NCT04758377
Title: Characterizing Hemorrhage in Acute Spinal Cord Injury With MRI
Acronym: CHASM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian Kwon, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H20-03585
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Traumatic Spinal Cord Haemorrhage
Keywords: vasopressors; magnetic resonance imaging
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Serial MRI scans of patients with acute cervical SCI to quantify hemorrhage.
  Interventions: Procedure: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Procedure: Magnetic resonance imaging (MRI) — Serial MRI scans of patients with acute cervical SCI to quantify hemorrhage.

SUMMARY:
The study is designed to determine whether hemorrhage within the injured spinal cord is influenced by mean arterial pressure (MAP) augmentation with vasopressors and by venous thromboembolism (VTE) prophylaxis with anticoagulants in the first two weeks following a traumatic spinal cord injury (tSCI).

DETAILED DESCRIPTION:
This will be a single-center prospective observational study of patients with an acute cervical traumatic spinal cord injury

ELIGIBILITY:
Inclusion Criteria:

* Acute tSCI injury involving bony spinal levels between C0 and T1
* Baseline Asia Impairment Scale (AIS) grade of A, B, or C
* Admission to study site within 24 hours of injury
* Male or female age 19 or older
* Able and willing to provide informed consent

Exclusion Criteria:

* Pathological fracture due to metabolic condition or neoplasia
* Spinal cord injury due to infection
* Presence of pacemaker, aneurysm clip or other device which is a contraindication to MRI
* BMI > 40 and unable to fit within the MRI scanner
* Multiple life threatening injuries (ISS >16) that make transport to MRI not in the patient's best interest
* Any condition that, at the time of admission, prevents a complete ISNCSCI assessment from being performed

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-02-06 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Hemorrhage Quantification 1 | Serial MRI assessments: Injury to 2 weeks post injury
  Area of hematoma
Hemorrhage Quantification 2 | Serial MRI assessments: Injury to 2 weeks post injury
  Vertical length of hematoma and vertical length of cord edema
Hemorrhage Quantification 3 | Serial MRI assessments: Injury to 2 weeks post injury
  The point of maximum cord compression vertebral level and anatomic point of maximum cord compression vertebral sublevel
Hemorrhage Quantification 4 | Serial MRI assessments: Injury to 2 weeks post injury
  Vertical length of cord edema rostral to maximum compression and vertical length of cord edema caudal to maximum compression.

SECONDARY OUTCOMES:
Hemodynamic Management Assessment 1 | Injury to 2 weeks post injury
  achieved mean arterial pressure
Hemodynamic Management Assessment 2 | Injury to 2 weeks post injury
  vasopressor usage/dose

OTHER OUTCOMES:
Neurologic Assessments | Injury to 6 months post injury
  International Standards for Neurological Classification of SCI (ISNCSCI)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kwon, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada